CLINICAL TRIAL: NCT01450995
Title: Open-label, 6 Month Crossover Study Evaluating Migraine Patient Satisfaction Comparing Treximet to 2 Aleve and 100mg Imitrex Taken Concomitantly
Brief Title: Migraine Treatment Satisfaction With Treximet Versus Concomitant 2 Aleve and Imitrex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stephen H. Landy, M.D. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Stephen H. Landy, M.D., Sponsor, Wesley Headache Clinic
Organization: Wesley Headache Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113403
Record Dates: First submitted 2011-09-02; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Migraine
Keywords: Migraine; Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — sumatriptan-naproxen; Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treximet (Active Comparator)
  Interventions: Drug: Treximet
- Imitrex and Aleve (Active Comparator)
  Interventions: Drug: Imitrex and two Aleve

INTERVENTIONS:
Drug: Treximet — Tablet form, one tablet dose, one tablet at migraine onset with second tablet for persistent or recurring migraine two hours after first dose.
  Arms: Treximet
Drug: Imitrex and two Aleve — Imitrex tablet, one tablet dose, Aleve tablets, 2 220 mg tablet dose. Three tablets taken concurrently with migraine onset. Second dose of tablets may be taken if migraine persists for two hours
  Arms: Imitrex and Aleve

SUMMARY:
This is an open label, 6 month cross over study in 50 migraine patients fulfilling International Headache Society Classification criteria for migraine headache with and without aura having 2-6 migraines per month and not over 14 days a month of headaches in the previous 3 months. Baseline Headache Impact Test -6 (HIT-6) will be obtained and 25 patients will administer Treximet as needed for 3 months and then 2 Aleve and 100mg Imitrex taken concomitantly as needed for 3 months. The other 25 patients will administer 2 Aleve and 100mg Imitrex taken concomitantly as needed for 3 months and then Treximet as needed for 3 months. In addition to Revised Patient Perception of Migraine Questionnaire (PPMQ-R)data, a detailed diary will be recorded regarding number of tablets taken per attack, compliance, rescue treatment, when patients treated their migraine attack (mild, moderate, or severe), onset of pain reduction (pain relief and pain free, and 24 hour pain relief and sustained pain free response.

DETAILED DESCRIPTION:
A migraine headache is characterized by pain felt on one and sometimes both side(s) of the head. Other symptoms associated with a migraine headache may include nausea, vomiting, and sensitivity to light and sound. A migraine can last a few hours or up to one or two days.

Triptan medications are currently thought to be safe and effective for acute migraine treatment. Treximet(tm) is a triptan tablet containing a combination of sumatriptan 85mg (Imitrex) and naproxen sodium 500 mg.

This combination has two methods of action for relieving a migraine headache. It targets the nerves and blood vessels involved in a migraine, and relieves inflammation that may cause migraine pain. Treximet(tm), is approved by the Food and Drug Administration.

The purpose of this research study is to compare the effectiveness of taking Treximet(tm) as a combination pill to taking two Aleve(r) tablets and 100mg of Imitrex(r) as separate tablets taken at the same time.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study if all of the following criteria apply:

1. Subject is male or female.
2. Subject is age 18 to 65.
3. A female is eligible to enter and participate in this study if she is not breast feeding and is of: non-childbearing potential (i.e. physiologically incapable of becoming pregnant) or child-bearing potential, has a negative urine pregnancy test at screening and agrees to use an acceptable method of contraception during the course of the study or, Female sterilization; or, Sterilization of male partner; or Implants of levonorgestrel; or Injectable progestogen; or Oral contraceptive (combined or progestogen only); or Any intrauterine device (IUD) meet this criterion; or Double barrier method; or Any other methods with published data showing that the lowest expected failure rate for that method is less than 1% per year
4. Subject has a diagnosis of migraine and meets IHS criteria for migraine with or without aura (1.1) or migraine with aura (1.2)
5. Subject has at least a 1-year history of migraine with 2-6 migraines per month in the three months prior to screening
6. Subject typically experiences moderate to severe migraine pain preceded by an identifiable mild pain phase.
7. Subject is able to read, understand and complete diaries, subject questionnaires and the instructions for the study.
8. Subject is able and willing to give written informed consent to participate in the study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subject has confirmed or suspected ischemic heart disease (angina pectoris, history of myocardial infarction, documented silent ischemia), Prinzmetal's angina, or signs/symptoms consistent with any of the above.
2. Subject has evidence or history of ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome.
3. Subject has cardiac arrhythmias requiring medication or a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study.
4. Subject has a history of cerebrovascular pathology including stroke.
5. Subject has a history of congenital heart disease.
6. Subject has uncontrolled hypertension at screening (sitting (>140 mmHg systolic pressure or >90mmHg diastolic pressure).
7. Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease.
8. Subject has significant peripheral vascular disease
9. Subject is currently taking any anti-coagulant (e.g., Coumadin®).
10. Subject has a history of inflammatory bowel disease.
11. Subject has a history of any bleeding disorder.
12. Subject has a history of GI ulceration in the past six months or gastrointestinal bleeding in the past year.
13. Subject is taking any antiplatelet agent (except low-dose aspiring ≤ 325 mg/day for cardioprotective reasons).
14. Subject is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker.
15. Subject has a history of epilepsy.
16. Subject has basilar migraine, hemiplegic migraine or cluster headache.
17. Subject has impaired renal, hepatic, of any gastrointestinal surgery, gastrointestinal obstruction or perforation.
18. Subject who is currently taking monoamine oxidase inhibitor drugs (MAOIs), or has taken any MAOI within 2 weeks prior to screening.
19. Subject is pregnant, actively trying to become pregnant or breast-feeding.
20. Subject has ≥ 15 headache days in any of the three previous months prior to screening.
21. Subject is of childbearing potential and not using adequate contraceptive measures.
22. Subject has evidence of a rebound headache pattern caused by ergotamines or analgesics in the past three months.
23. Subject has evidence of alcohol or substance abuse within the last year, which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results.
24. Subject has any concurrent medical condition which may affect the interpretation of efficacy and safety data or which otherwise contraindicates participation in this clinical trial.
25. Subject has participated in an investigational drug trial within the previous four weeks, or plans to participate in another study at any time during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Measurement of patient satisfaction of Treximet vs 2 Aleve and 100mg Imitrex | one year

SECONDARY OUTCOMES:
Measurement of time to onset of pain relief | One year
Measurement of time to onset of pain free | one year
Measurement of 24 hour sustained pain free | One year
Measurement of 24 hour sustained pain relief | One year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Landy, M.D., Principal Investigator — Wesley Headache Clinic
Locations (1):
- Wesley Headache Clinic, Memphis, Tennessee, United States

REFERENCES:
- [Result] Revicki DA, Kimel M, Beusterien K, Kwong JW, Varner JA, Ames MH, Mahajan S, Cady RK. Validation of the revised Patient Perception of Migraine Questionnaire: measuring satisfaction with acute migraine treatment. Headache. 2006 Feb;46(2):240-52. doi: 10.1111/j.1526-4610.2006.00289.x. PMID 16492233
- [Result] Landy S, DeRossett SE, Rapoport A, Rothrock J, Ames MH, McDonald SA, Burch SP. Two double-blind, multicenter, randomized, placebo-controlled, single-dose studies of sumatriptan/naproxen sodium in the acute treatment of migraine: function, productivity, and satisfaction outcomes. MedGenMed. 2007 Jun 7;9(2):53. PMID 17955107
- [Result] Smith T, Blumenthal H, Diamond M, Mauskop A, Ames M, McDonald S, Lener S, Burch S. Sumatriptan/Naproxen sodium for migraine: efficacy, health related quality of life, and satisfaction outcomes. Headache. 2007 May;47(5):683-92. doi: 10.1111/j.1526-4610.2007.00790.x. PMID 17501849
- [Result] 4. Cady RK, et al. Consistent medication satisfaction with sumatriptan RT Technology and naproxen sodium for acute migraine treatment. Poster presented at 13th Congress of the International Headache Society (IHS), June 28-July 1, 2007; Stockholm, Sweden.
- [Result] Mathew NT, Landy S, Stark S, Tietjen GE, Derosier FJ, White J, Lener SE, Bukenya D. Fixed-dose sumatriptan and naproxen in poor responders to triptans with a short half-life. Headache. 2009 Jul;49(7):971-82. doi: 10.1111/j.1526-4610.2009.01458.x. Epub 2009 May 27. PMID 19486178
- [Result] Kimel M, Hsieh R, McCormack J, Burch SP, Revicki DA. Validation of the revised Patient Perception of Migraine Questionnaire (PPMQ-R): measuring satisfaction with acute migraine treatment in clinical trials. Cephalalgia. 2008 May;28(5):510-23. doi: 10.1111/j.1468-2982.2007.01524.x. Epub 2008 Mar 31. PMID 18384420